CLINICAL TRIAL: NCT03990662
Title: Predictors of Good Outcomes Following Manual Therapy in Patients With Temporomandibular Disorders: Development and Validation Studies
Brief Title: What Are the Clinical Factors Associated With a Significant Pain Reduction Following Physiotherapy in Patients With Temporomandibular Disorders?
Status: Completed | Type: Observational
Sponsor: Istituto Stomatologico Italiano (Other)
Collaborators: University of Birmingham (Other)
Responsible Party: Principal Investigator, Giacomo Asquini, Physiotherapist at the Italian Stomatologic Institute - Craniomandibular Physiotherapy Service, Istituto Stomatologico Italiano
Other Study IDs: PredictorsOutcomeTMD2019GA
Record Dates: First submitted 2019-06-17; First posted 2019-06-19 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Temporomandibular Disorders
Keywords: Temporomandibular Joint Dysfunction Syndrome; Manual Therapy; Prediction; Pain
MeSH Terms: conditions — Temporomandibular Joint Disorders; Temporomandibular Joint Dysfunction Syndrome; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- TMD: Patients (aged ≥18 years) with a diagnosis of Temporomandibular Disorders
  Interventions: Other: Physiotherapy - Manual Therapy

INTERVENTIONS:
Other: Physiotherapy - Manual Therapy — Participants will receive four sessions of manual therapy applied to craniomandibular structures over four weeks. The application of manual therapy aims to decrease pain by treating masticatory muscle trigger points, muscle tightness, and restricted temporomandibular joint movements. Several techniques will be considered, including ventral and caudal anterior glide temporomandibular joint mobilisation, soft tissue interventions for the management of trigger points in masticatory muscles and myofascial induction therapy applied to craniomandibular structures. The structures targeted in the treatment sessions will be the temporomandibular joint, temporal muscles, masseter muscles, medial and lateral pterygoid muscles and suprahyoid muscles.

SUMMARY:
RATIONALE OF THE OBSERVATION STUDY:

This study aims to observe which patients with temporomandibular disorder improve more following a physiotherapy program of four sessions. Knowing the characteristics of patients who have the most significant improvements could help clinician advise or advise against physiotherapy for the treatment of temporomandibular disorders.

STUDY PROCEDURES The study will be conducted at the Istituto Stomatologico Italiano. Patients diagnosed with Temporomandibular Disorder will be recruited in the gnathological and neuromuscular gnathological departments. The physiotherapists of the Craniomandibular Physiotherapy Service will perform physiotherapy therapy, which consists of four physiotherapy sessions [lasting 30 minutes, about once a week] over a month. Before starting the treatment, participants will be asked to answer some questions concerning their state of health (e.g. pain intensity) with particular reference to Temporomandibular Disorder (e.g. location and duration of pain). The intensity of pain and the level of function will then be monitored at baseline, after 4 weeks and after 8 weeks from baseline.

EXPECTED BENEFITS FROM THE STUDY AND EXPECTED BENEFITS FOR THE PATIENT The benefits are the discovery of new knowledge in the field of therapeutic choice for patients with temporomandibular disorder.

DETAILED DESCRIPTION:
Additional information:

In this study protocol, the variables reported in the section "Other Pre-specified Outcomes" are the predictors that will be included in the prediction model.

The total "Enrollment" is 180 participants (100 for the development phase and 80 for the validation phase).

ELIGIBILITY:
Inclusion Criteria:

* (1) adults aged ≥18 years;
* (2) TMD diagnosis according to the Axis I of the Diagnostic Criteria for TMDs (DC/TMD) (Shiffman et al., 2014);
* (3) no therapeutic interventions reported (for their TMD) in the past six months (Wahlund et al., 2015);
* (4) capacity to use and understand written and verbal Italian language;
* (5) mental capacity to provide informed consent.

Exclusion Criteria:

* (1) TMD pain related to rheumatoid/inflammatory arthritis;
* (2) any physical or mental condition that could potentially influence the study;
* (3) they commence another treatment for their TMD (pharmacology, oral appliance, others) throughout the duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited in a Dental Hospital [TMJ Unit].
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2019-06-14 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Change in Pain Intensity (Visual Analogue Scale [VAS]) from baseline to one month | Change from baseline to one month
  Pain intensity will be calculated by averaging the ratings of current pain, average pain in the past week, and worst pain in the past week using the Visual Analogue Scale (VAS), consisting of a horizontal line measuring 10 cm (without marks), with "no pain" written at the left extremity, and "worst pain imaginable" at the right extremity. Patients will be educated to trace a perpendicular line on the horizontal line to intend the pain intensity. The distance from the 0 points will be after measured in millimetres. The VAS is a reliable and valid scale to assess pain intensity as an outcome measure in intervention studies. Based on the Initiative on Methods, Measurement, and Pain Assessment in Clinical Trials (IMMPACT) recommendations about TMD , a reduction of at least 30% of the VAS score for pain intensity is considered clinically significant. Consequently, a reduction in the total VAS score [≥ 30%] will be defined as a good outcome
Change in Pain Intensity (Visual Analogue Scale [VAS]) from baseline to two month | Change from baseline to two month
  Pain intensity will be calculated by averaging the ratings of current pain, average pain in the past week, and worst pain in the past week using the Visual Analogue Scale (VAS), consisting of a horizontal line measuring 10 cm (without marks), with "no pain" written at the left extremity, and "worst pain imaginable" at the right extremity. Patients will be educated to trace a perpendicular line on the horizontal line to intend the pain intensity. The distance from the 0 points will be after measured in millimetres. The VAS is a reliable and valid scale to assess pain intensity as an outcome measure in intervention studies. Based on the Initiative on Methods, Measurement, and Pain Assessment in Clinical Trials (IMMPACT) recommendations about TMD , a reduction of at least 30% of the VAS score for pain intensity is considered clinically significant. Consequently, a reduction in the total VAS score [≥ 30%] will be defined as a good outcome
Change in Function (patient specific functional scale [PSFS]) from baseline to one month | Change from baseline to one month
  To capture a potential change in function, patients will also complete the patient specific functional scale (PSFS). The PSFS is a self reported outcome measure assessing functional change in patients with musculoskeletal disorders. It is responsive to clinically significant change over time, even in chronic pain patients. Patients are invited to rate, on an 11-point scale, their level of difficulty performing at least three different daily activities. Following the treatment, patients are required to score again the activities previously rated. It is known the PSFS is a valid, reliable, and responsive outcome measure with a high test-retest reliability in patients with lower back pain and knee problems.
Change in Function (patient specific functional scale [PSFS]) from baseline to two month | Change from baseline to two month
  To capture a potential change in function, patients will also complete the patient specific functional scale (PSFS). The PSFS is a self reported outcome measure assessing functional change in patients with musculoskeletal disorders. It is responsive to clinically significant change over time, even in chronic pain patients. Patients are invited to rate, on an 11-point scale, their level of difficulty performing at least three different daily activities. Following the treatment, patients are required to score again the activities previously rated. It is known the PSFS is a valid, reliable, and responsive outcome measure with a high test-retest reliability in patients with lower back pain and knee problems.

OTHER OUTCOMES:
Pain during maximal mouth opening | Baseline, one month, two months
  Pain intensity during maximal mouth opening will be measured via a Numeric Rating Scale (NRS) . Participants will be asked: "Rate your pain by indicating the number that best describes pain during maximal mouth opening, with 0 meaning 'No pain' and '10' meaning 'Pain as bad as you can imagine' " . NRS is a reliable and valid tool to detect pain modification in clinical trials.
Central sensitisation: Central Sensitisation Inventory (CSI) | Baseline
  Participants will be asked to complete the Italian version of the CSI. CSI examines existing health symptoms through a 0-100 score for 25 items, each with five alternatives from 'never' (score 0) to 'always' (score 4). The CSI has adequate test-retest reliability and internal consistency in people with and without pain. The Italian version of the CSI has an acceptable Cronbach's alpha [0.87]
Treatment expectations | Baseline
  Participants will report if they "Completely disagree", "Somewhat disagree", "Neutral", "Somewhat agree", "Completely agree" with the following statement: "I believe that manual techniques applied to my jaw will significantly help to improve my pain". Only answers "somewhat agree" or "completely agree" are considered positive treatment expectations.
Duration of TMD pain | Baseline
  The duration of TMD pain will be collected in days and obtained from open hospital records and patient interviews
Maximal mouth opening (MMO) | Basiline, one month, two months
  MMO measurements will be in millimetres and calculated with a ruler in a neutral craniocervical position (e.g., sitting or supine) as suggested by the DC/TMD. The measurement procedure follows the DC/TMD protocol. MMO in a neutral craniocervical position is a reliable clinical measures and has good inter and intra-rater reliability
Number of pain locations | Baseline
  Participants will complete a pain drawing representing spatial pain distribution through a body frontal and dorsal view chart. The pain reported in distinct body regions (e.g., head, jaw area, back area, pelvic area, neck area) will be collected as the number of painful sites

CONTACTS AND LOCATIONS:
Overall Officials: Giacomo Asquini, Principal Investigator — Istituto Stomatologico Italiano
Locations (1):
- Istituto Stomatologico Italiano, Miano, Milano, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Asquini G, Devecchi V, Borromeo G, Tessera P, Russillo A, Michelotti A, Bucci R, Falla D. External Validation of a Clinical Prediction Tool for the Use of Manual Therapy in Patients With Temporomandibular Disorders. J Oral Rehabil. 2026 Feb;53(2):515-528. doi: 10.1111/joor.70092. Epub 2025 Nov 11. PMID 41216702
- [Derived] Asquini G, Devecchi V, Edoardo Bianchi A, Borromeo G, Tessera P, Falla D. External validation of a clinical prediction tool for the use of manual therapy for patients with temporomandibular disorders: a protocol for a prospective observational study. BMJ Open. 2023 Jul 14;13(7):e069327. doi: 10.1136/bmjopen-2022-069327. PMID 37451727
- [Derived] Asquini G, Devecchi V, Borromeo G, Viscuso D, Morato F, Locatelli M, Falla D. Predictors of pain reduction following a program of manual therapies for patients with temporomandibular disorders: A prospective observational study. Musculoskelet Sci Pract. 2022 Dec;62:102634. doi: 10.1016/j.msksp.2022.102634. Epub 2022 Jul 31. PMID 35939919
- [Derived] Asquini G, Bianchi AE, Borromeo G, Locatelli M, Falla D. The impact of Covid-19-related distress on general health, oral behaviour, psychosocial features, disability and pain intensity in a cohort of Italian patients with temporomandibular disorders. PLoS One. 2021 Feb 2;16(2):e0245999. doi: 10.1371/journal.pone.0245999. eCollection 2021. PMID 33529226
- [Derived] Asquini G, Bianchi AE, Heneghan NR, Rushton AB, Borromeo G, Locatelli M, Falla D. Predictors of pain reduction following manual therapy in patients with temporomandibular disorders: a protocol for a prospective observational study. BMJ Open. 2019 Nov 12;9(11):e032113. doi: 10.1136/bmjopen-2019-032113. PMID 31722951